CLINICAL TRIAL: NCT02923622
Title: Efficacy and Safety Evaluation of Traditional Chinese Medicine in the Treatment of Advanced Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Sponsor
Other Study IDs: D161100005116002
Record Dates: First submitted 2016-09-23; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Advanced Colorectal Cancer; Traditional Chinese Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Traditional Chinese and Western medicine combined group
  Interventions: Other: Integrated traditional Chinese and Western medicine
- Traditional Chinese medicine group
  Interventions: Other: Traditional Chinese medicine herbals
- Western medicine group
  Interventions: Other: Western medicine

INTERVENTIONS:
Other: Traditional Chinese medicine herbals — TCM herbal treatment based on TCM syndrome differentiation，without any anti tumor therapy in Western Medicine
  Groups: Traditional Chinese medicine group
Other: Integrated traditional Chinese and Western medicine — TCM herbal treatment combine with anti tumor therapy in Western Medicine ( including non recommended chemotherapy, radiotherapy and targeted therapy in clinical guidelines)
  Groups: Traditional Chinese and Western medicine combined group
Other: Western medicine — Anti tumor therapy in Western Medicine ( including non recommended chemotherapy, radiotherapy and targeted therapy in clinical guidelines)
  Groups: Western medicine group

SUMMARY:
Although patients of colorectal cancer use Traditional Chinese Medicine (TCM) herbal therapy extensively in China, no strong evidence exists to demonstrate the safety and survival outcomes of TCM herbal therapy combined with conventional western medicine for treatment of this disease. The purpose of this multi-center perspective cohort study is to evaluate the relationship between TCM herbal therapy and survival outcomes in patients with advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed adenocarcinoma of the colon or rectum
* TNM classification of stage IV disease according to American Joint Committee on Cancer
* Between 18 and 80 years old
* Progression or inability undergone conventional chemotherapy (Conventional chemotherapy regimen containing fluorouracil, oxaliplatin, irinotecan based chemotherapy, and all the above regimen should be used before)
* Expected survival time is over 3 months
* Signed informed consent

Exclusion Criteria:

* serious non-malignant diseases such as heart, renal, and hepatic illnesses
* the presence of other types of malignancies
* The patients can not take medicine for intestinal obstruction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients with advanced colorectal cancer and the tumor progressed after conventional chemotherapy
Sampling Method: Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
Progress free survival | 3 years
Quality of life as assessed by FACT-C v4.0 | 3 years
Tumor control rate | 3 years
TCM syndrome score | 3 years
Number of participants with treatment-related adverse events as assessed by Chinese version of CTCAE v4.0 | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Department of Xiyuan hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hao TT, Xu Y, Cui N, Qu Q, Liang BY, Yuan JH, Zhao Y, Li QN, Lu F, Wu Y. Effectiveness and Safety Evaluation of Chinese Medicine in Treatment of Metastatic Colorectal Cancer after Chemotherapy Failure: Protocol of a Prospective Multicenter Cohort Study. Chin J Integr Med. 2021 Sep;27(9):674-679. doi: 10.1007/s11655-020-3420-0. Epub 2020 Aug 19. PMID 32820453